CLINICAL TRIAL: NCT04655963
Title: Neuromodulation and Plasticity in Cognitive Control Neurocircuitry in Chronic Stroke
Brief Title: Brain Stimulation for Improving Cognition in Chronic Stroke (NEPTUNE)
Acronym: NEPTUNE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00083136; 3P2CHD086844-04S1 (NIH)
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Stroke
Keywords: stroke; rTMS; cognition
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All participants would receive open-label treatment for approximately eight, 3-minute sessions of intermittent theta burst rTMS on each of three days within a seven-day span.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dose 1 (Experimental): All participants would receive open-label treatment for approximately eight, 3-minute sessions of intermittent theta burst rTMS on each of three days within a seven-day span. A single session=600 pulses at 120% rMT, iTBS triplets at 50 Hz for 2 s and repeated every 10 s for a total of 190 s to left dlPFC. Total pulses=14,400.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — MagVenture MagPro TMS System would be utilized to deliver 3-minute sessions of intermittent theta burst to left dorsolateral prefrontal cortex.

SUMMARY:
Few treatments are available for post-stroke rehabilitation. The current study aims to develop a novel, short-term, high-dose repetitive transcranial magnetic stimulation (rTMS) based intervention to improve post-stroke cognitive problems. This study will test the safety as well as changes in cognitive function and brain activation with the administration of an accelerated rTMS protocol in chronic stroke.

DETAILED DESCRIPTION:
The goal of this pilot study is to determine whether a repetitive high-dose form of non-invasive brain stimulation is a promising and safe treatment for stroke-related cognitive difficulties. Repetitive transcranial magnetic stimulation (rTMS) is an FDA approved treatment for depression, and is used commonly to treat people for their depression. In studies of rTMS for depression and other disorders, individuals have experienced improved cognitive function. Thus, we are testing here whether cognitive function in individuals with chronic stroke could be improved by rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Have right hemisphere ischemic or hemorrhagic stroke within last 6 months chronicity
* Able to perform given cognitive tasks
* No metal implanted in the body
* A negative urine pregnancy test, if female subject of childbearing potential.

Exclusion Criteria:

* Primary intracerebral hematoma or subarachnoid hemorrhage
* Bi-hemispheric ischemic strokes
* Other concomitant neurological disorders affecting motor or cognitive function
* History of seizure disorder
* Preexisting scalp lesion or wound or bone defect or hemicraniectomy
* Substance use disorder
* Psychotic disorders
* Claustrophobia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Side Effects as assessed by iTBS Review of Systems | Approximately 6 months.
  This study will be demonstrating the safety of using rTMS in stroke patients by assessing adverse events and side effects using the intermittent transcranial brain stimulation (iTBS) Review of Systems questionnaire. The minimum value of the iTBS scale is 0 and the maximum is 75, the higher the score the more severe the side effects meaning a worse outcome.
Assess feasibility, of an accelerated protocol of rTMS in stroke patients looking at retention and using an rTMS a credibility questionnaire pre/post treatment. | Approximately 6 months.
  This study will be demonstrating the feasibility of using rapid transcranial magnetic stimulation (rTMS) in stroke patients by assessing retention throughout the study and using a credibility scale. The credibility scale maximum is 36 and minimum is 0, a higher ratings means higher credibility score which is a better outcome.
Demonstrate acceptability of an accelerated protocol of rTMS in stroke patients using an acceptability of rTMS questionnaire. | Approximately 6 months.
  This study will be demonstrating the acceptability of using rapid transcranial magnetic stimulation (rTMS) in stroke patients by using an rTMS acceptability scale. The acceptability scale maximum is 100 and the minimum is 0, a higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-03-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT04655963/ICF_002.pdf